CLINICAL TRIAL: NCT02443194
Title: The Effect of Duloxetine on Mood, Quality of Life and Cognitive Functioning in Glioblastoma Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: principle investigator decision due to many adverse events in patients
Sponsor: michal roll (Other Government)
Responsible Party: Sponsor-Investigator, michal roll, Director R & D, Tel-Aviv Sourasky Medical Center
Organization: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0124-15 TLV
Record Dates: First submitted 2015-05-03; First posted 2015-05-13 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Depression
Keywords: depression; glioblastoma
MeSH Terms: conditions — Depression; Glioblastoma | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group # 1- ACTIVE (Active Comparator): Patients who underwent resection or biopsy of glioblastoma (newly diagnosed glioblastoma), will randomization ratio of 1: 1 by the pharmacist (by age, KPS, the degree of tumor resection) two research groups:
  Group # 1: consisting of 50 patients who will be treated immediately after diagnosis, 30 mg Cymbalta duloxetine -morning for a week and then a dose exceeding 60 mg for 3 months.
  Interventions: Drug: duloxetine
- Group # 2-PLACEBO (Placebo Comparator): Group # 2 will include 50 patients treated immediately after diagnosis with placebo for 3 months
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: duloxetine — after randomization the patient will receive cymbalta/ placebo for 3 months
  Other Names: cymbalta
  Arms: Group # 1- ACTIVE
Drug: PLACEBO — after randomization the patient will receive cymbalta/ placebo for 3 months
  Arms: Group # 2-PLACEBO

SUMMARY:
Primary tumor glioblastoma is the most common malignant brain. Standard treatment includes biopsy or excision of the tumor in order to obtain a pathological diagnosis, and tumor mass reduction. After the surgery patients are treated with radiation and Temodal. The most common psychiatric symptom in this patient population is depression, valued at up to approximately 50% in patients with glioma . Depression not only adversely affects the quality of life of patients but also impairs the ability and cognitive function due to the complex clinical course of patients with glioblastoma. There is a tendency to give Diagnosis of depression in this patient population, due to a lack of awareness, knowledge and literature on the subject. This study was designed to prospectively randomized, controlled, double-blind study.

This method of recruitment - patients who undergo resection or biopsy of glioblastoma (newly diagnosed glioblastoma), immediately after diagnosis, patients will receive an explanation about the study and sign a consent form will enter research.

DETAILED DESCRIPTION:
This study was designed to prospectively randomized, controlled, double-blind study.This method of recruitment patients who undergo resection or biopsy of glioblastoma (newly diagnosed glioblastoma), immediately after diagnosis, patients will receive an explanation about the study and sign a consent form will enter research.

Patients who underwent resection or biopsy of glioblastoma (newly diagnosed glioblastoma), will randomization ratio of 1: 1 by the pharmacist (by age, Karnofsky score, the degree of tumor resection) two research groups:

Group # 1: consisting of 50 patients who will be treated immediately after diagnosis, 30 mg Cymbalta morning for a week and then a dose exceeding 60 mg for 3 months.

Group # 2: will include 50 patients treated immediately after diagnosis placebo for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who signed an informed consent form
* Patients who underwent resection or biopsy for GBM
* KPS> 70

Exclusion Criteria:

* Patients being treated with antidepressants
* Unable to answer the questionnaires because of an inability to communicate
* Patients being treated; monoamine oxidase inhibitors (MAOI) CYP1A2 Inhibitors or (CYP2D6 inhibitors (SSRIs such as fluoxetine, paroxetine, or anti-arrhythmia such as quinidine) Patients with Glaucoma, narrow angle
* Severe renal dysfunction. According to laboratory criteria specified earlier.
* Hepatic insufficiency - which laboratory criteria mentioned earlier.
* Pregnant women Patients Dementia
* Patients who previously suffered from depression in the past or within 5 years of diagnosis, and currently do not receive drug therapy
* Sensitivity to any of its ingredients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
changes in patients mood and cognitive function according to the neuropsychological assessment | 3 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Grossman, MD, Principal Investigator — Neurosurgery department, Tel Aviv Medical Center

REFERENCES:
- [Result] Greer TL, Sunderajan P, Grannemann BD, Kurian BT, Trivedi MH. Does duloxetine improve cognitive function independently of its antidepressant effect in patients with major depressive disorder and subjective reports of cognitive dysfunction? Depress Res Treat. 2014;2014:627863. doi: 10.1155/2014/627863. Epub 2014 Jan 19. PMID 24563781